CLINICAL TRIAL: NCT01420484
Title: Noninvasive Blood Pressure Measuring
Brief Title: CNAP in Heart Surgery
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Collaborators: CNSystems Medizintechnik AG (Industry)
Responsible Party: Principal Investigator, Konstanze Plaschke, PhD, Heidelberg University
Other Study IDs: S234/2009
Record Dates: First submitted 2011-08-18; First posted 2011-08-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Transfemoral Implantation of Aortic Valves
Keywords: CNAP; continuous non-invasive arterial pressure; IAP; blood pressure; analgosedation; high-risk patients; rapid-pacing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- different blood pressure intervals
  Interventions: Other: different blood pressure intervals

INTERVENTIONS:
Other: different blood pressure intervals — In differnent blood presure intervals the IAP and CNAP measurement differences will be observed.

SUMMARY:
The role of continuous non-invasive arterial pressure (CNAP) in high risk patients with pronounced variation of arterial pressure will be assessed under analgosedation.

Therefore, patients will be analyzed during normo-, hypo- and hypertension with standard IAP undergoing elective transfemoral aortic valve implantation procedures. Systolic, diastolic, and mean invasive arterial pressures (IAP) will be compared to those obtained by CNAP. Data will be analysed in different periods of arterial pressure for agreement of the two methods and for determination of precision (i.e. measurement error) and accuracy (i.e. systematic error). Additionally, we will compare both methods regarding the amplitude and time of very fast changes in arterial pressure during intervals of functional cardiac arrests (rapid pacing).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for elective transfemoral implantation of the aortic valve in analgosedation will be included.
* The patients' primary diagnosis was severe aortic stenosis, that was defined as a valve area of <1cm² or a mean pressure gradient >50mmHg.

Exclusion Criteria:

* an advanced dysfunction of peripheral perfusion (i.e. pronounced arterial peripheral artery occlusive disease or Raynaud's syndrome)
* arterio-venous shunts for haemodialysis, and vascular surgery of the upper extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted for elective transfemoral implantation of the aortic valve in analgosedation will be included. The patients' primary diagnosis was severe aortic stenosis, that was defined as a valve area of <1cm² or a mean pressure gradient >50mmHg.
  Exclusion criteria for the study will be an advanced dysfunction of peripheral perfusion (i.e. pronounced arterial peripheral artery occlusive disease or Raynaud's syndrome), arterio-venous shunts for haemodialysis, and vascular surgery of the upper extremities.
  Before including patients in the present study, blood pressure will be measured on both arms noninvasively by oscillometry to exclude any significant arterial stenosis between the upper extremities. Differences of less than 10 mmHg will be accepted.
  All patients won't receive any sedative drugs preoperatively and were allowed to drink fluids up to 2 hours before surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
blood pressure | blood pressure

SECONDARY OUTCOMES:
age | age
  descriptive data

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schramm, MD, Principal Investigator — Department of Anesthesiology
Locations (1):
- Medical Clinic, University of heidelberg, Heidelberg, Germany